CLINICAL TRIAL: NCT02374489
Title: A Phase II Trial of LDK378 as the First or Second-line Therapy in ROS1 and /or ALK Over-expressed Advanced Intrahepatic or Hilar Cholangiocarcinoma
Brief Title: A Phase II Trial of LDK378 in ROS1 and /or ALK Over-expressed Advanced Intrahepatic or Hilar Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: ROS1 in IHC and gene rearrangement result can not match。No tumor response。
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T3214
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-01

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm studies (Experimental): LDK378 in suitable patients:
  Collect tumor tissue for immunohistochemistry staining to confirm the status of ROS1 or ALK expression. If the patient fits all criteria, LDK378 750 mg ( p.o.) daily, with 3 week as a treatment cycle
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378 — LDK378 750 mg ( p.o.) daily, with 3 week as a treatment cycle.
  Other Names: ceritinib(Zykadia)

SUMMARY:
Primary objective:

To investigate the objective response rate in patients with ROS1 or ALK over-expressed locally advanced, or metastatic intrahepatic or hilar cholangiocarcinoma receiving LDK378 Secondary objectives:The progression-free survival ,The disease control rate ,The overall survival ,The toxicity profiles , The correlation between clinical outcomes and the potential predictive biomarker for tumor response

DETAILED DESCRIPTION:
Sample size: LDK378 will be considered as an active agent and deserved for further development. Considering 10% dropout rate, total 34 patients will be included.

Step 1: LDK378 in suitable patients:

Collect tumor tissue for immunohistochemistry staining to confirm the status of ROS1 or ALK expression. If the patient fits all criteria, LDK378 750 mg ( p.o.) daily, with 3 week as a treatment cycle.

Step 2: Evaluation of tumor response according to RECIST 1.1 version

1. Evaluation will be done at baseline and every 6 weeks
2. Evaluation will be performed with CT or MRI and the response is defined as follows:

   * Complete response - the disappearance of all target lesions.
   * Partial response - at least a 30% decrease in the sum of the longest diameter of target lesions compared to the baseline sum longest diameter.
   * Progressive disease - at least a 20% increase in the sum of the longest diameter of target lesions compared to the smallest sum longest diameter recorded since the treatment started or the appearance of one, or more new lesions, or reappearance of any lesion that had disappeared, or clear worsening of any assessable disease, or appearance of any new lesion or site.
   * Stable disease - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, compared to the smallest sum longest diameter since the treatment started

ELIGIBILITY:
Inclusion Criteria:

* 1.Histological or cytologically confirmed diagnosis of intrahepatic or hilar cholangiocarcinoma that demonstrates ALK and/or ROS1 over-expression by IHC (3+).
* 2.Locally advanced with inoperable or metastatic disease status
* 3.ECOG performance status 0-2.
* 4.Aged no less than 20 years and no more than 75 years, at the time of acquisition of informed consent 5.Patients must have recovered from all toxicities related to prior anticancer therapies to ≤ grade 2 (CTCAE v 4.03), provided that concomitant medication is given prior to initiation of treatment with LDK378. Exception to this criterion: patients with any grade of alopecia are allowed to enter the treatment.

  6.The following laboratory criteria have been met:

  •Absolute neutrophil count (ANC) ≥1.5 x 109/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥ 75 x 109/L
  * Serum total bilirubin ≤1.5 x upper limit of normal (ULN), except for patients with biliary tract obstruction statis post drainage or stent may be included if total bilirubin ≤3.0 x ULN and direct bilirubin≤ 1.5 x ULN
  * Aspartate transaminase (AST) < 3.0 x ULN, except for patients with liver metastasis, who are only included if AST < 5 x ULN; alanine transaminase (ALT) < 3.0 x ULN, except for patients with liver metastasis, who are only included if ALT < 5 x ULN
  * Calculated or measured creatinine clearance (CrCL) ≥ 30 mL/min 7.Patient must have the following laboratory values or have the following laboratory values corrected with supplements to be within normal limits at screening:
  * Potassium ≥ 1.0 x lower limit of normal (LLN)
  * Magnesium ≥ 1.0 x LLN
  * Phosphorus ≥ 1.0 x LLN
  * Total calcium (corrected for serum albumin) ≥ 1.0 x LLN 8.At least one, not previously irradiated, measurable lesion according to RECIST (version 1.1) 9.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

* 1.Patients with known hypersensitivity to any of the excipients of LDK378 (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate).

  2.Patients with symptomatic CNS metastases who are neurologically unstable or have required increasing doses of steroids within the 1 week prior to study entry to manage CNS symptoms.

  3.Prior therapy with LDK378. 4.Other anti-tumor agent such as systemic chemotherapy, immunotherapy or targeted therapy within 2 weeks before the commencement of study treatment.

  5.Presence or history of a malignant disease other than cholangiocarcinoma that has been diagnosed and/or required therapy within the past year and is not undergoing active anticancer treatment. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.

  6.Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention).

  7.Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:unstable angina within 6 months prior to screening;myocardial infarction within 6 months prior to screening;history of documented congestive heart failure (New York Heart Association functional classification III-IV);uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication ;initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;ventricular arrhythmias; supraventricular and nodal arrhythmias not controlled with medication;other cardiac arrhythmia not controlled with medication;corrected QTc (male: QTc >450 msec; female: QTc> 470 msec ) using Bazett correction on the screening ECG.

  8.Impaired GI function or GI disease that may alter absorption of LDK378 or inability to swallow up to five LDK378 capsules daily.

  9.Ongoing GI adverse events > grade 2 (e.g. nausea, vomiting, or diarrhea) at the start of the study.

  10.Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with LDK378 and for the duration of participation:Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes .Strong inhibitors or strong inducers of CYP3A4/5 ;Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, CYP2C8 and/or CYP2C9 ;Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (eg, dabigatran, rivaroxaban, apixaban).;increasing doses of corticosteroids;enzyme-inducing anticonvulsive agents;herbal supplements 11.Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

  12.Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after the last dose of study treatment. Highly effective contraception methods include:Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.

Male sterilization (at least 6 months prior to screening) with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. For female subjects on the study the vasectomized male partner should be the sole partner for that subject.

Combination of any two of the following (a+b or a+c or b+c):

1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

13.Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after the last dose of study treatment. Male patients for 3 months should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
objective response rate | three year
  Evaluation of tumor response according to RECIST 1.1 version

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Cheng Kung University Hospital, Taipei